CLINICAL TRIAL: NCT00140764
Title: Intravaginal Treatment of Disturbances of Vaginal Flora Among HIV Infected and Uninfected Women in Malawi
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: METRO STUDY
Record Dates: First submitted 2005-08-30; First posted 2005-09-01 (Estimated); Last update posted 2011-08-10 (Estimated); Status verified 2011-08

CONDITIONS: Bacterial Vaginosis; Trichomonas Vaginitis; Urogenital Diseases
Keywords: Genitourinary symptoms
MeSH Terms: conditions — Vaginosis, Bacterial; Trichomonas Vaginitis; Urogenital Diseases

INTERVENTIONS:
Drug: Metronidazole gel versus placebo gel

SUMMARY:
The purpose of this intervention is to find out whether intravaginal treatment with a gel containing an antibiotic (metronidazole), compared to a similar placebo gel (without antibiotic), can reduce the frequency of bacterial vaginosis, a common vaginal infection among African women who are HIV uninfected or HIV infected. The study will also determine the effect of these vaginal gels on genitourinary symptoms.

DETAILED DESCRIPTION:
This is a phase 3, randomized, double masked, two arms study conducted in Malawi, Southeast Africa. The study is conducted among nonpregnant HIV infected or uninfected women of reproductive age. Intermittent mass treatment approaches are followed where women are randomized to antibiotic intravaginal treatment or placebo at enrollment. Women receive assigned product every three months for one year.

ELIGIBILITY:
Inclusion Criteria:

Nonpregnant HIV-Uninfected HIV-Infected

Exclusion Criteria:

Pregnant

Ages: 18 Years to 55 Years | Sex: Female
Age Groups: Adult
Dates: Start 2003-01; Study Completion 2005-03

PRIMARY OUTCOMES:
Prevalence of bacterial vaginosis
Reported genitourinary symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Taha E Taha, MD PHD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health

REFERENCES:
- [Derived] Aizire J, Dadabhai S, Taulo F, Makanani B, Gadama L, Sun J, Tsui A, Taha TE. Use of effective family planning methods and frequency of sex among HIV-infected and HIV-uninfected African women. Contracept Reprod Med. 2018 Jul 9;3:10. doi: 10.1186/s40834-018-0063-z. eCollection 2018. PMID 30002871